CLINICAL TRIAL: NCT05229432
Title: Pilot Assessment to Find Evidence of Gastric Motility Abnormalities in Eosinophilic Gastric Disorders
Brief Title: Study of Gastric Motility in Eosinophilic Gastritis
Acronym: OAT-FEED
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0349
Record Dates: First submitted 2021-12-20; First posted 2022-02-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Gastritis; Gastroparesis; Gastric Motility Disorder
Keywords: Gastritis; Eosinophilic Gastrointestinal Disorders; Gastric Dysfunction; Gastric Dysmotility; Eosinophils; Eosinophilia; Eosinophilic Disorders; Digestive System Diseases; Immune System Diseases; Stomach Diseases; Gastric Emptying Scintigraphy; Endoscopy
MeSH Terms: conditions — Eosinophilic enteropathy; Gastroparesis; Gastritis; Eosinophilic Esophagitis; Eosinophilia; Digestive System Diseases; Immune System Diseases; Stomach Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Purpose:

The study is a cross-sectional observational study designed to determine if eosinophilic gastritis (EG) results in gastric motility impairment.

Hypothesis:

Gastric dysfunction occurs in the natural history of EG but is underdiagnosed due, in part, to contraindications to the use of the standard meals used in gastric emptying studies.

ELIGIBILITY:
Inclusion Criteria:

* Eosinophilic gastritis (EG) defined as at least one endoscopy with histopathologic evidence of ≥ 30 eosinophils in 5 or more high powered fields (hpf's) with associated symptoms of EG.
* Patient reported symptoms starting at least one year or more prior to screening consistent with a diagnosis of EG: nausea, vomiting, early satiety, abdominal pain/bloating, regurgitation, diarrhea.
* Symptoms suggestive of a possible gastric motility disorder during the 60 days prior to screening including: nausea, vomiting, early satiety, post-prandial feeling of fullness or bloating.
* Tolerance and willingness to consume the oatmeal meal in this study.

Exclusion Criteria:

* Diagnosis of eosinophilic enteritis.
* Inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
* Known disorders associated with eosinophilic gastrointestinal (GI) diseases (e.g., D 816 V Kit+ systemic mastocytosis, Marfan syndrome or Loey's Dietz Syndrome).
* Known inflammatory or autoimmune disorders associated with gastric dysmotility such as systemic sclerosis, lupus or eosinophilic fasciitis.
* Uncontrolled diabetes or known diabetic complications of gastroparesis, neuropathy or nephropathy.
* Taking opioid agents in the 2 weeks prior to screening and throughout the study.
* History of strictures in the small bowel or stomach (e.g., pyloric stenosis) or gastric surgeries or procedures such as pyloromyotomy, pyloric dilation, pyloric resection, vagotomy, bariatric surgery or post-Nissen fundoplication or antrectomy with Billroth I, Billroth II or Roux-en-Y gastrojejunostomy.
* Past or current medical problems or findings such as: advanced liver disease (Child's B or C), acute or chronic renal disease (serum creatinine > 3 mg/dL), neurologic disease (e.g., dysautonomia), achalasia and adrenal insufficiency.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males and females aged 18 and 59 years old with EG.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gastric motility disorders determined via gastric emptying scintigraphy (GES) imaging at timepoints 0 minutes, 30 minutes, 60 minutes, 120 minutes and 180 minutes (% of meal remaining/time). | Gastric Emptying Scintigraphy [0 minutes, 30 minutes, 60 minutes, 120 minutes and 180 minutes]
  A gastric motility disorder will be defined as the presence of delayed gastric emptying ( > 8% of an oatmeal meal remaining in the stomach at 3 hours) measured by gastric emptying scintigraphy (GES).
  Specifically, the participant will consume oatmeal with a small amount of mixed-in radioactive material. After consuming the meal, a gastric emptying scintigraphy scan will take images at the following timepoints: 0 minutes, 30 minutes, 60 minutes, 120 minutes and 180 minutes.

SECONDARY OUTCOMES:
Relationship between gastric dysfunction and eosinophilic gastritis disease activity measured via peak and mean eosinophils/hpf in the stomach. | Endoscopy Procedure (Peak and mean eosinophils/hpf [Date of GES + 2-10 days])
  The relationship between gastric dysfunction and eosinophilic gastritis disease activity, as represented by eosinophil levels, will be measured via the correlation between the time it takes the oatmeal to leave the stomach and the amount of eosinophils that the pathologists count in pieces of tissue (biopsies) from the stomach obtained during the endoscopy procedure.
  The higher the number of eosinophils in the tissue, the more active the EG disease is considered to be.
Relationship between gastric dysfunction and eosinophilic gastritis disease activity measured via symptomology and quality of life questionnaires. | Questionnaires [screening/baseline visit, 2 weeks prior to date of GES up to completion of the endoscopy]
  The correlation between the time it takes the oatmeal to leave the stomach and patient-reported data on the following questionnaires: 'Patient Assessment of Gastrointestinal Symptom Severity Index' (PAG-SYM), 'Patient Assessment of Gastrointestinal Quality of Life' (PAGI-QoL), 'Patient Reported Outcome Measurement Information System' (PROMIS) and 'Symptoms of Eosinophilic Gastritis' (EoG-SQ).
  PAG-SYM: 20 items each with a 6-point Likert scale ranging from 0="None'' to 5="Very Severe''. Higher scores are associated with more severe symptoms.
  PAGI-QoL: 30 items each with a 6-point Likert scale ranging from 0="None of the time'' to 5="All of the time''. A higher score means a higher quality of life.
  PROMIS: 29 items each with a 5-point Likert scale. A higher score represents a worse quality of life.
  EoG-SQ: the severity of EG symptoms on a scale of 0 to 10. The frequency of symptoms on a scale of 0 to 7. Higher scores indicate a greater symptom burden.
Relationship between gastric dysfunction and eosinophilic gastritis disease activity measured via assessing endoscopic features of the stomach. | Endoscopy Procedure (Endoscopic features [Date of GES + 2-10 days])
  The relationship between gastric dysfunction and eosinophilic gastritis disease activity measured via endoscopic features utilizing the 'Eosinophilic Gastritis Endoscopy Score' (EoG-REFS). During the endoscopy, the physician will look at the stomach and record what it looks like on the EoG-REFS assessment.
  EoG-REFS scoring: Utilizes standardized criteria for the presence and degree of 5 major endoscopic features (granularity, nodularity, erosion/ulceration, friability, erythema). Total score is the maximum score of the 5 feature scores from the body, antrum or fundus. Total scores range from 0 - 14. Higher scores indicate more severe endoscopic findings. There is also a 'Global Assessment of Endoscopic Severity' with a scale from 0 (normal) to 10 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Paneez Khoury, MD, Study Chair — National Institutes of Health (NIH)
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - The National Institutes of Health, Bethesda, Maryland
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No